CLINICAL TRIAL: NCT06037616
Title: Comparison of Methods for Teaching Simple Skin Sutures to Medical Students: a Randomized Blinded Controlled Study
Brief Title: Teaching Simple Skin Sutures to Medical Students
Acronym: E-SUTURE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023 LAUTRETTE E-SUTURE
Record Dates: First submitted 2023-08-30; First posted 2023-09-14 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-08

CONDITIONS: Medical Students

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- gr A: powerpoint and tutor (Active Comparator): teaching with powerpoint and tutor
  Interventions: Other: powerpoint and tutor
- gr B: powerpoint and tutor and video skill (Active Comparator): teaching with powerpoint and tutor and video showing skill to perform a skin suture
  Interventions: Other: powerpoint and tutor; Other: video skill
- gr C: powerpoint and tutor and video error (Active Comparator): teaching with powerpoint and tutor and video showing errors
  Interventions: Other: powerpoint and tutor; Other: video errors
- gr D: powerpoint and tutor and video skill and error (Active Comparator): teaching with powerpoint and tutor and video showing skill to perform a skin suture and errors
  Interventions: Other: powerpoint and tutor; Other: video skill; Other: video errors

INTERVENTIONS:
Other: powerpoint and tutor — Powerpoint on indication of skin suture and tutor for the skill to perform skin suture
Other: video skill — Video showing skill to perform a skin suture
  Arms: gr B: powerpoint and tutor and video skill; gr D: powerpoint and tutor and video skill and error
Other: video errors — Video showing errors of skin suture
  Arms: gr C: powerpoint and tutor and video error; gr D: powerpoint and tutor and video skill and error

SUMMARY:
Learning the simple skin suture is part of the surgical basics required for all medical students, including future general practitioners.

However, there is no data in the educational literature to help choose the best learning technique.

Several teams have offered video learning showing the correct technique. Level n+1 peer learning was also proposed, without and with supervision by an expert.

The investigators propose to carry out a prospective study comparing the quality of sutures and knowledge according to the chosen learning method.

DETAILED DESCRIPTION:
Send to medical student a teaching package two weeks before simulation session to practice skin suture. There are 4 teaching packages related to 4 interventional groups The skin suture performed by medical students are recorded on video. 1 video per medical student.

The skin sutures recorded in these video are rated by two blinded expert with evaluation grid.

After the simulation session, the students complete knowledge, self-confidence, satisfaction and mental load questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Medical student of the faculty of Clermont-Ferrand

Exclusion Criteria:

* Refusal to participate

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
quality of skin suture | 15 days after simulation session
  Quality of suture on anonymized video recording during the assessment day, rated by the blinded expert using an evaluation grid evaluation grid is made up of 14 items from the litterature the minimum value is: 0 (worse outcome) and maximum value is: 15 points (better outcome)

SECONDARY OUTCOMES:
knowledge of student | 15 days after simulation session
  8 multiple choice questions (5 items per MCQ); the minimum value is: 0 (worse outcome) and maximum value is: 8 points (better outcome)
self-confidence of student | 15 days after simulation session
  self evaluation with a Likert scale (5points); point 0 corresponds to "no confidence"; point 5 corresponds to "total confidence"
mental load of student | 15 days after simulation session
  self evaluation with a Likert scale (9points); point 0 corresponds to "very low"; point 9 corresponds to "very high"

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Lautrette, Principal Investigator — CHU de Clermont-Ferrand; Nicolas D'Ostrevy, Principal Investigator — CHU de Clermont-Ferrand; geraud galvaing, Principal Investigator — Centre Jean Perrin
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France